CLINICAL TRIAL: NCT03397979
Title: Twice Daily Versus Twice Weekly Soak-and-Seal Baths in Pediatric Atopic Dermatitis: A Randomized, Single-blinded, Prospective Crossover Controlled Trial
Brief Title: Twice Daily Versus Twice Weekly Soak-and-Seal Baths in Pediatric Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Ivan Cardona, Clinical Assistant Professor, Tufts University School of Medicine, MaineHealth
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3927
Record Dates: First submitted 2017-09-28; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; bathing; baths
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Randomized, Single-blinded, Prospective Crossover Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A single treating physician assessed outcomes and, along with those analyzing the data, was masked to group assignment. In other words, the care provider, investigator, and outcomes assessor were blinded to which bathing arm (twice daily or twice weekly) the study participants were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrequent soaking baths (Active Comparator): Infrequent soaking baths, in this study, is defined as twice a week soaking baths for 10 minutes or less, over 2 weeks. However, this is a crossover study design with two interventions: 1) Infrequent soaking baths, as defined above, and 2) Frequent soaking baths (defined as twice daily soaking baths for 15-20 minutes, over 2 weeks). All subjects in the study will undergo both interventions, but in different order. Thus, this is a study comparing Infrequent Versus Frequent Soaking Baths. Each subject serves as their own control.
  Interventions: Behavioral: Infrequent versus Frequent Soaking Baths
- Frequent soaking baths (Active Comparator): Frequent soaking baths, in this study, is defined as twice daily soaking baths for 15-20 minutes, over 2 weeks. However, this is a crossover study design with two interventions: 1) Infrequent soaking baths, as defined in the first arm description above, and 2) Frequent soaking baths, as defined above in this arm description. All subjects in the study will undergo both interventions, but in different order. Thus, this is a study comparing Infrequent Versus Frequent Soaking Baths. Each subject serves as their own control.
  Interventions: Behavioral: Infrequent versus Frequent Soaking Baths

INTERVENTIONS:
Behavioral: Infrequent versus Frequent Soaking Baths — Submersion of skin, affected by atopic dermatitis, in a bathtub filled with luke-warm water, where the frequency and duration of these baths are varied, to look for any differential effect.
  Other Names: Soak and seal baths; Soak and smear baths

SUMMARY:
There are few studies evaluating best bathing practices in the management of pediatric atopic dermatitis (AD). Trans-epidermal water loss plays a key role in the pathophysiology of AD. In concert with application of topical corticosteroids (TCS), we sought to investigate whether frequent soaking baths (i.e. twice daily for two weeks), followed immediately by application of an occlusive moisturizer (i.e. soak-and-seal), would be more effective than infrequent soaking baths (i.e. twice weekly for two weeks) in the management of AD.

DETAILED DESCRIPTION:
To evaluate the effectiveness of twice daily soak-and-seal baths for improving severity of disease in children with AD, we implemented a randomized clinical trial using a single-blind, crossover-controlled design. Patients received the same moisturizer, cleanser, and class VI topical corticosteroid (TCS), and only bathing varied. After a 1 week run-in, children were randomized 1:1 into 2 groups: Group 1 underwent twice weekly soak-and-seal baths for 2 weeks ("dry method") followed by twice daily soak-and-seal baths for 2 weeks ("wet method"), and group 2 did the converse. A single treating physician assessed outcomes and, along with those analyzing the data, was masked to group assignment. Participants and their caregivers could not be masked. Analyses were based on intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children ages 6 months to 11 years of age with moderate to severe atopic dermatitis according to the criteria of Hanifin and Rajka.

Exclusion Criteria:

* Patients with suspected or established primary immune deficiency, patients receiving systemic corticosteroids, ultraviolet light therapy, immuno-therapeutic agents, and/or anti-infective drugs less than 1 month from the onset of the study.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2011-11-14 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
SCORAD (SCORing Atopic Dermatitis eczema severity score) | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion criteria. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in SCORAD from baseline (V2), for visits 3 minus visits 4.
  SCORAD (which stands for SCORing Atopic Dermatitis eczema severity score) is a validated eczema severity score assessed by the treating physician. The scale ranges from 0-103, with higher numbers correlating with more severe/worse eczema.

SECONDARY OUTCOMES:
ADQ (Atopic Dermatitis Quickscore eczema severity score) | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion criteria. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in ADQ from baseline (V2), for visits 3 minus visits 4.
  ADQ (which stands for Atopic Dermatitis Quickscore) is a validated eczema severity score assessed by the caregivers of a child with AD. The scale ranges from 0-70, with higher numbers correlating with more severe/worse eczema.
IDQOL (Infant Dermatitis Quality of life index for under 4 years of age) | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion criteria. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in IDQOL from baseline (V2), for visits 3 minus visits 4.
  IDQOL (Which stands for Infant Dermatitis Quality of life index) is a validated quality of life measuring tool for AD. The scale ranges from 0-44, with higher numbers correlating with more severe/worse eczema.
CDLQI (Children's Dermatology Life Quality Index for 4 years of age and older) | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion criteria. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in CDLQI from baseline (V2), for visits 3 minus visits 4.
  CDLQI (Which stands for Children's Dermatology Life Quality Index) is a validated quality of life measuring tool for AD. The scale ranges from 0-40, with higher numbers correlating with more severe/worse eczema.
DFI (Dermatitis Family Impact questionnaire for QOL measure for 5 and up) | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion criteria. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in DFI from baseline (V2), for visits 3 minus visits 4.
  DFI (which stands for Dermatitis Family Impact) is a validated quality of life measuring tool for AD. The scale ranges from 0-40, with higher numbers correlating with more severe/worse eczema.
Staphylococcal aureus (S. aureus); relative quantities | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in S. aureus from baseline (V2), for visits 3 minus visits visits 4.
  Relative quantities of S. aureus cultured from the skin. The scale ranges from 1+ rare, 2+ few, 3+ moderate, 4+ many, with higher numbers correlating with higher quantities of S. aureus on the skin.
Skin hydration status | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in skin hydration from baseline (V2), for visits 3 minus visits 4.
  Skin hydration status as measured by impedance-based capacitance utilizing the DPM 9003 instrument by Nova Tech. Corp. The scale ranges from 90-999, with higher values correlating with greater skin hydration.
Amount of topical corticosteroid (Desonide 0.05% Oint.) used | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in Desonide use from baseline (V2), for visits 3 minus visits 4.
  Amount of Desonide 0.05% Oint. used based on weighing the desonide tube at each visit
Amount of topical moisturizer (Vanicream) used | Each subject undergoes 4 visits over 5 weeks. Visit 1 (V1) to establish if subject fulfills inclusion. V2 (baseline) is after a 1 week "run-in". 2 weeks between V2-V3 and V3-V4. Change in Vanicream use from baseline (V2), for visits 3 minus visits 4.
  Amount of Vanicream used based on weighing the Vanicream container at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Ivan D Cardona, M.D., Principal Investigator — Allergy & Asthma Associates of Maine
Locations (1):
- Allergy and Asthma Associates of Maine, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No
Able to share any and all individual participant data with other researchers if asked.

REFERENCES:
- [Background] Bieber T. Atopic dermatitis. N Engl J Med. 2008 Apr 3;358(14):1483-94. doi: 10.1056/NEJMra074081. No abstract available. PMID 18385500
- [Background] Elias PM, Hatano Y, Williams ML. Basis for the barrier abnormality in atopic dermatitis: outside-inside-outside pathogenic mechanisms. J Allergy Clin Immunol. 2008 Jun;121(6):1337-43. doi: 10.1016/j.jaci.2008.01.022. Epub 2008 Mar 7. PMID 18329087
- [Background] Akdis CA, Akdis M, Bieber T, Bindslev-Jensen C, Boguniewicz M, Eigenmann P, Hamid Q, Kapp A, Leung DY, Lipozencic J, Luger TA, Muraro A, Novak N, Platts-Mills TA, Rosenwasser L, Scheynius A, Simons FE, Spergel J, Turjanmaa K, Wahn U, Weidinger S, Werfel T, Zuberbier T; European Academy of Allergology and Clinical Immunology/American Academy of Allergy, Asthma and Immunology. Diagnosis and treatment of atopic dermatitis in children and adults: European Academy of Allergology and Clinical Immunology/American Academy of Allergy, Asthma and Immunology/PRACTALL Consensus Report. J Allergy Clin Immunol. 2006 Jul;118(1):152-69. doi: 10.1016/j.jaci.2006.03.045. PMID 16815151
- [Background] Sator PG, Schmidt JB, Honigsmann H. Comparison of epidermal hydration and skin surface lipids in healthy individuals and in patients with atopic dermatitis. J Am Acad Dermatol. 2003 Mar;48(3):352-8. doi: 10.1067/mjd.2003.105. PMID 12637914
- [Background] Cork MJ, Robinson DA, Vasilopoulos Y, Ferguson A, Moustafa M, MacGowan A, Duff GW, Ward SJ, Tazi-Ahnini R. New perspectives on epidermal barrier dysfunction in atopic dermatitis: gene-environment interactions. J Allergy Clin Immunol. 2006 Jul;118(1):3-21; quiz 22-3. doi: 10.1016/j.jaci.2006.04.042. Epub 2006 Jun 9. PMID 16815133
- [Background] Werner Y, Lindberg M. Transepidermal water loss in dry and clinically normal skin in patients with atopic dermatitis. Acta Derm Venereol. 1985;65(2):102-5. PMID 2408409
- [Background] Chandar P, Nole G, Johnson AW. Understanding natural moisturizing mechanisms: implications for moisturizer technology. Cutis. 2009 Jul;84(1 Suppl):2-15. PMID 19702109
- [Background] O'Regan GM, Sandilands A, McLean WHI, Irvine AD. Filaggrin in atopic dermatitis. J Allergy Clin Immunol. 2008 Oct;122(4):689-693. doi: 10.1016/j.jaci.2008.08.002. Epub 2008 Sep 5. PMID 18774165
- [Background] McLean WH, Palmer CN, Henderson J, Kabesch M, Weidinger S, Irvine AD. Filaggrin variants confer susceptibility to asthma. J Allergy Clin Immunol. 2008 May;121(5):1294-5; author reply 1295-6. doi: 10.1016/j.jaci.2008.02.039. Epub 2008 Apr 8. No abstract available. PMID 18395783
- [Background] Tilles G, Wallach D, Taieb A. Topical therapy of atopic dermatitis: controversies from Hippocrates to topical immunomodulators. J Am Acad Dermatol. 2007 Feb;56(2):295-301. doi: 10.1016/j.jaad.2006.09.030. PMID 17224373
- [Background] Burkhart CG. Clinical assessment by atopic dermatitis patients of response to reduced soap bathing: pilot study. Int J Dermatol. 2008 Nov;47(11):1216-7. doi: 10.1111/j.1365-4632.2008.03829.x. No abstract available. PMID 18986472
- [Background] Hanifin JM, Tofte SJ. Update on therapy of atopic dermatitis. J Allergy Clin Immunol. 1999 Sep;104(3 Pt 2):S123-5. doi: 10.1016/s0091-6749(99)70054-0. PMID 10482863
- [Background] Tarr A, Iheanacho I. Should we use bath emollients for atopic eczema? BMJ. 2009 Nov 13;339:b4273. doi: 10.1136/bmj.b4273. No abstract available. PMID 19914950
- [Background] Gutman AB, Kligman AM, Sciacca J, James WD. Soak and smear: a standard technique revisited. Arch Dermatol. 2005 Dec;141(12):1556-9. doi: 10.1001/archderm.141.12.1556. PMID 16365257
- [Background] Chiang C, Eichenfield LF. Quantitative assessment of combination bathing and moisturizing regimens on skin hydration in atopic dermatitis. Pediatr Dermatol. 2009 May-Jun;26(3):273-8. doi: 10.1111/j.1525-1470.2009.00911.x. PMID 19706087
- [Background] Kameyoshi Y, Tanaka T, Mochizuki M, Koro O, Mihara S, Hiragun T, Tanaka M, Hide M. [Taking showers at school is beneficial for children with severer atopic dermatitis]. Arerugi. 2008 Feb;57(2):130-7. Japanese. PMID 18349587
- [Background] Mochizuki H, Muramatsu R, Tadaki H, Mizuno T, Arakawa H, Morikawa A. Effects of skin care with shower therapy on children with atopic dermatitis in elementary schools. Pediatr Dermatol. 2009 Mar-Apr;26(2):223-5. doi: 10.1111/j.1525-1470.2009.00887.x. PMID 19419481
- [Background] Cardona ID, Cho SH, Leung DY. Role of bacterial superantigens in atopic dermatitis : implications for future therapeutic strategies. Am J Clin Dermatol. 2006;7(5):273-9. doi: 10.2165/00128071-200607050-00001. PMID 17007538
- [Background] Huang JT, Abrams M, Tlougan B, Rademaker A, Paller AS. Treatment of Staphylococcus aureus colonization in atopic dermatitis decreases disease severity. Pediatrics. 2009 May;123(5):e808-14. doi: 10.1542/peds.2008-2217. PMID 19403473
- [Background] Breneman DL, Hanifin JM, Berge CA, Keswick BH, Neumann PB. The effect of antibacterial soap with 1.5% triclocarban on Staphylococcus aureus in patients with atopic dermatitis. Cutis. 2000 Oct;66(4):296-300. PMID 11109156
- [Background] Kubota K, Machida I, Tamura K, Take H, Kurabayashi H, Akiba T, Tamura J. Treatment of refractory cases of atopic dermatitis with acidic hot-spring bathing. Acta Derm Venereol. 1997 Nov;77(6):452-4. doi: 10.2340/0001555577452454. PMID 9394980
- [Background] Murota H, Takahashi A, Nishioka M, Matsui S, Terao M, Kitaba S, Katayama I. Showering reduces atopic dermatitis in elementary school students. Eur J Dermatol. 2010 May-Jun;20(3):410-1. doi: 10.1684/ejd.2010.0928. Epub 2010 Apr 23. No abstract available. PMID 20413368
- [Background] Schuttelaar ML, Coenraads PJ. A randomized, double-blind study to assess the efficacy of addition of tetracycline to triamcinolone acetonide in the treatment of moderate to severe atopic dermatitis. J Eur Acad Dermatol Venereol. 2008 Sep;22(9):1076-82. doi: 10.1111/j.1468-3083.2008.02716.x. Epub 2008 Apr 1. PMID 18384552
- [Background] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Background] Carel K, Bratton DL, Miyazawa N, Gyorkos E, Kelsay K, Bender B, Strand M, Atkins D, Gelfand EW, Klinnert MD. The Atopic Dermatitis Quickscore (ADQ): validation of a new parent-administered atopic dermatitis scoring tool. Ann Allergy Asthma Immunol. 2008 Nov;101(5):500-7. doi: 10.1016/S1081-1206(10)60289-X. PMID 19055204
- [Background] Lewis-Jones MS, Finlay AY, Dykes PJ. The Infants' Dermatitis Quality of Life Index. Br J Dermatol. 2001 Jan;144(1):104-10. doi: 10.1046/j.1365-2133.2001.03960.x. PMID 11167690
- [Background] 27. Hanifin JM, Rajka G. Diagnostic features of atopic derma titis. Acta Derm Venereol1980;92:44-7.
- [Background] Woo SI, Kim JY, Lee YJ, Kim NS, Hahn YS. Effect of Lactobacillus sakei supplementation in children with atopic eczema-dermatitis syndrome. Ann Allergy Asthma Immunol. 2010 Apr;104(4):343-8. doi: 10.1016/j.anai.2010.01.020. PMID 20408346
- [Background] Gruber C, Wendt M, Sulser C, Lau S, Kulig M, Wahn U, Werfel T, Niggemann B. Randomized, placebo-controlled trial of Lactobacillus rhamnosus GG as treatment of atopic dermatitis in infancy. Allergy. 2007 Nov;62(11):1270-6. doi: 10.1111/j.1398-9995.2007.01543.x. PMID 17919141
- [Background] Meggitt SJ, Gray JC, Reynolds NJ. Azathioprine dosed by thiopurine methyltransferase activity for moderate-to-severe atopic eczema: a double-blind, randomised controlled trial. Lancet. 2006 Mar 11;367(9513):839-46. doi: 10.1016/S0140-6736(06)68340-2. PMID 16530578